CLINICAL TRIAL: NCT03042728
Title: Impact of Inclusion of a Dog as Part of the Fibromyalgia Treatment Program on Patient's Physical and Mental Health Functioning - A Randomized Controlled Trial
Brief Title: Impact of Inclusion of a Therapy Dog Visit as Part of the Fibromyalgia Treatment Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Arya B. Mohabbat, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-006296
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dog interaction (Active Comparator): Dog interaction will be received by patients in addition to usual care of fibromyalgia.
  Interventions: Behavioral: Dog Interaction
- Human Interaction (Active Comparator): Human interaction will be received by patients in addition to usual care of fibromyalgia.
  Interventions: Behavioral: Human Interaction

INTERVENTIONS:
Behavioral: Dog Interaction — A therapy dog will visit the patients.
  Arms: Dog interaction
Behavioral: Human Interaction — A human will visit the patients.
  Arms: Human Interaction

SUMMARY:
In this study the investigators hypothesize that the presence of a Mayo Clinic certified therapy dog will provide additional benefits above typical therapy for patients suffering from fibromyalgia currently enrolled in the Mayo Clinic Fibromyalgia Program.

DETAILED DESCRIPTION:
The human animal bond refers an emotional relationship between animals and people. The purpose of this study is to evaluate whether the presence of a dog provide additional benefits above typical therapy for patients suffering from fibromyalgia and also to assess the emotional wellbeing state of the therapy dog.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with Fibromyalgia at our Fibromyalgia Clinic
* Patients actively being seen at the Fibromyalgia Clinic
* Able and willing to give informed consent
* Able to speak English
* Able to complete questionnaires
* No fear or allergy of dogs

Exclusion Criteria

* Diagnoses of bipolar disorder, schizophrenia, or dementia
* Individuals who decline to participate in the study
* Individuals that are severely allergic to or fearful of dogs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Revised Fibromyalgia Impact Questionnaire (FIQR) score | Baseline to 1.5 day
  The FIQR questionnaire consists of 21 questions in 3 domains. Each question has 11 boxes similar to a visual analog scale, rating the item from no difficulty to very difficult. To score the FIQR, the researcher must sum the answers for each domain. Then the function domain is divided by 3, the overall impact domain remains unchanged, and the symptom domain score is divided by 2. The resulting scores are added, and final score can range from 0 -100, with 0=no difficulty, and 100=great difficulty.

SECONDARY OUTCOMES:
Change in Pain Intensity Score (Numeric Rating Scale (NRS)) | Baseline to 1.5 day
  The subject is asked to make three pain ratings corresponding to the current, best, and worst pain experienced over the past 24 hours. The average of the 3 ratings is used to represent the patient's level of pain over the previous 24 hours. The NRS scale consists of numbers 0 through 10, with 0=no pain, 1-3=mild pain, 4-6=moderate pain, and 7-10=severe pain.
Change in Score for Fatigue, Anxiety, and Depression | Baseline to 1.5 day
  The subject is asked to rate their symptoms on a visual analog scale from 1-10, with 1=not at all, and 10=unbearable.

CONTACTS AND LOCATIONS:
Overall Officials: Arya B Mohabbat, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes